CLINICAL TRIAL: NCT04727437
Title: STOPping Anticoagulation for Isolated or Incidental Subsegmental Pulmonary Embolism
Acronym: STOPAPE
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Birmingham (Other)
Collaborators: Royal United Hospitals Bath NHS Foundation Trust (Other); Cimar (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Worktribe 799297; 280586 (Other: IRAS); ISRCTN15645679 (Other: ISRCTN)
Record Dates: First submitted 2021-01-07; First posted 2021-01-27 (Actual); Last update posted 2021-09-29 (Actual); Status verified 2021-09

CONDITIONS: Subsegmental Pulmonary Embolism Nos
MeSH Terms: interventions — Warfarin; N(4)-oleylcytosine arabinoside; Heparin, Low-Molecular-Weight

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (Active Comparator): Full dose anticoagulation treatment as standard care for at least 3 months.
  Interventions: Drug: Warfarin; Drug: direct oral anticoagulants; Drug: Low molecular weight heparin
- Intervention (Experimental): Withholding anticoagulation for Isolated Sub-Segmental Pulmonary Embolism (ISSPE) for at least 3 months.
  Interventions: Other: No treatment

INTERVENTIONS:
Other: No treatment — Withholding anticoagulation for at least 3 months.
  Arms: Intervention
Drug: Warfarin — anticoagulation drug given for at least 3 months.
  Arms: Control
Drug: direct oral anticoagulants — anticoagulation drug given for at least 3 months.
  Arms: Control
Drug: Low molecular weight heparin — anticoagulation drug, subcutaneous injection given for at least 3 months.
  Arms: Control

SUMMARY:
Pulmonary embolisms (PE) occur when blood clots cause a blockage of the blood supply to the lungs. A small PE located in the subsegmental pulmonary vasculature is identified as a subsegmental PE (SSPE). Anticoagulants are used to treat SSPE and work by preventing new clots from forming whilst the body's own mechanisms break down the clots, however they can also increase the risk of major and potentially life threatening bleeding. More recent observational data of routine care for SSPE showed very high complication rates of anticoagulation but in patients where treatment was withheld, this proved to be a safe strategy in terms of recurrent venous thromboembolism (VTE).

Computed tomography pulmonary angiography (CTPA) scans are now able to detect SSPE, however there are concerns that there is an over-diagnosis due to the incorrect interpretation of small artefacts. 1466 patients from approximately 50 sites will be recruited, these sites will consist of hospitals across the United Kingdom (UK). Patients 18 and over with isolated SSPE, confirmed by either CTPA or CT thorax with IV contrast, will be eligible for the trial. Patients will be randomised to either receive standard anticoagulation for at least 3 months (control) or no anticoagulation for at least 3 months (intervention). The participant will receive telephone follow up calls at 4, 12 and 24 weeks following the end of their treatment, and additional data will also be taken from their medical records at these time points. The participant isn't required to be contacted for the 52 week follow up as the data will be extracted from the National Health Service (NHS) Digital collection of Hospital Episode Statistics (HES). In total participation in the study will last 12 months. In addition the cost-effectiveness of no treatment versus treatment with full anticoagulation will be looked at and also improving on radiological diagnosis of SSPE.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years
* SSPE diagnosed by the radiologist at the trial site by CTPA or CT thorax with IV contrast
* No evidence of proximal deep vein thrombosis on doppler ultrasonography or CT / Magnetic Resonance venography
* Heart rate (<110bpm)
* Systolic blood pressure (≥100 mmHg)
* Oxygen saturation (≥90%)
* Written signed informed consent to the trial

Exclusion Criteria:

* Indication for hospital admission
* >7 days empirical anticoagulation treatment immediately prior to randomisation
* <28 days since first symptoms of proven or clinically suspected Coronavirus disease (COVID-19)
* Known stage 5 chronic kidney disease
* Patients with active cancer defined as cancer diagnosed within the past 6 months, cancer for which anticancer treatment was being given at the time of enrolment or during 6 months before randomisation, or recurrent locally advanced or metastatic cancer
* Patients with previous unprovoked PE, thrombophilia or requiring long term anticoagulation for another reason
* Patients with a Deep Vein Thrombosis / thrombus of an unusual site (e.g. upper limbs, associated with a line) that requires anticoagulation
* Patients with active bleeding
* Any condition which, in the opinion of the investigator, makes the participant unsuitable for trial entry due to prognosis/terminal illness with a projected survival of less than 3 months
* Pregnancy confirmed by positive pregnancy test or post-partum period or actively trying to conceive
* Inability to comply with the trial schedule and follow-up
* Participation in a Clinical Trial of Investigative Medicinal Product (CTIMP) study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1466 (Estimated)
Dates: Start 2021-04-08 (Actual); Primary Completion 2023-07 (Estimated); Study Completion 2024-05 (Estimated)

PRIMARY OUTCOMES:
A composite score of the number of recurrent venous thromboembolism and/or clinically relevant bleeding | 3 months
  To determine if withholding anticoagulation is non-inferior to standard anticoagulation therapy in the treatment of isolated or incidental subsegmental pulmonary embolism for preventing recurrent venous thromboembolism, and/or death related and non death related venous thromboembolism, or superior for clinically relevant bleeding over 3 months, compared with at least 3 months of full anticoagulation. This will be measured using a scoring system which is currently being developed by the statistical team, and will be detailed in the statistical analysis plan when finalised.

SECONDARY OUTCOMES:
The change in frequency and severity of harmful events | 6 and 12 months
  Determine whether withholding anticoagulation for isolated subsegmental pulmonary embolism reduces harmful events (recurrent venous thromboembolism, clinically relevant bleeding) compared with at least 3 months of full anticoagulation at 6 and 12 months. This will be assessed through Hospital Episode Statistic records.
Number of new diagnosis of pulmonary hypertension of right ventricular dysfunction identified from Hospital Episode Statistics. | 12 months
  Determine the impact of withholding anticoagulation for isolated subsegmental pulmonary embolism on diagnoses of pulmonary hypertension at 12 months. Measure new diagnosis of pulmonary hypertension or right ventricular dysfunction within 12 months of subsegmental pulmonary embolism, defined from Hospital Episode Statistics clinical coding and supported where possible by additional radiological data and echocardiogram undertaken in tertiary pulmonary hypertension centres. The parameters and variables used to analysed data from the Hospital Episode Statistics are being developed and will be outlined in the statistical analysis plan when finalised.
Reclassification rate from thoracic radiologist review | 32 months
  Determine the reclassification rate of subsegmental pulmonary embolism diagnoses made by acute reporting radiologists when reviewed by thoracic radiologists and formulate a set of rules to improve acute reporting radiologists' diagnoses of subsegmental pulmonary embolism.
Measuring the rate of net clinical benefit | 3 and 6 months
  A composite of clinically relevant bleeding and recurrent venous thromboembolism at 3 and 6 months, measured at the 3 and 6 month follow up time points using statistical coding as described in the statistical analysis plan.
Measuring the rate of mortality | 3, 6 and 12 months
  Measurement of all-cause mortality and venous thromboembolism related mortality at 3, 6 and 12 months. Measurement of cardiovascular mortality at 3, 6 and 12 months defined as cardiac deaths (e.g. cardiogenic shock, fatal arrhythmia, cardiac rupture) and vascular deaths (e.g. venous thromboembolism related, fatal stroke, ruptured aortic aneurysm, aortic dissection).

OTHER OUTCOMES:
Healthcare resource use and cost | 12 months
  An economic evaluation will be undertaken to assess the cost-effectiveness of no treatment versus full dose anticoagulation in patients with isolated or incidental subsegmental pulmonary embolism. The base-case evaluation will take the form of an incremental cost-utility analysis to estimate cost per quality adjusted life year (QALY) over a 24 week follow up period using a version of the EuroQol descriptive questionnaire (EQ-5 Dimensions -5Levels), and a cost-effectiveness analysis to estimate cost per venous thromboembolism avoided over 52 weeks using routine data sources. Both analyses will be from a health services perspective. Additional analysis, using decision modelling, will explore the cost utility and cost-effectiveness of a pragmatic treatment policy (without expert thoracic radiological review) over a 52 week time horizon.
Behavioural analysis of the participants | 32 months
  To determine whether not treating subsegmental pulmonary embolism is acceptable to patients. To determine the health seeking behaviours and health utilisation of a no anticoagulation treatment strategy for isolated or incidental subsegmental pulmonary embolism. Selected patients will be interviewed by the qualitative researchers using a pre-set interview schedule via telephone or video calls.
Behavioural analysis of the healthcare professionals | 32 months
  To determine whether not treating subsegmental pulmonary embolism is acceptable to healthcare professionals. To determine the health seeking behaviours and health utilisation of a no anticoagulation treatment strategy for isolated subsegmental pulmonary embolism. Selected healthcare professionals will be interviewed by the qualitative researchers using a pre-set interview schedule via telephone or video calls.

CONTACTS AND LOCATIONS:
Locations (1):
- Surrey & Sussex Healthcare NHS Trust, Redhill, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes